CLINICAL TRIAL: NCT01988376
Title: Comparing the Rate of Insufficient Cells for Diagnosis Between Surepath® and Conventional Smear in Women After Radiation Therapy for Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 100140-E
Record Dates: First submitted 2013-08-16; First posted 2013-11-20 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2015-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

ARMS (2):
- Women with cervical cancer receive Surepath for screening (Experimental): Women will receive Surepath as a tool for screening the recurrence of cervical cancer.
  Interventions: Device: Surepath
- Women receive conventional Pap smear for screening (Active Comparator): Women who will receive conventional Pap smear for screening
  Interventions: Device: Conventional Pap smear

INTERVENTIONS:
Device: Surepath — A liquid-base method of Pap smear for screening the recurrence of cervical cancer
  Arms: Women with cervical cancer receive Surepath for screening
Device: Conventional Pap smear — Conventional Pap smear
  Arms: Women receive conventional Pap smear for screening

SUMMARY:
Background/Purpose: This is a large scale, multicenter randomized clinical trial to assess the feasibility of using SurePath® in cervical cancer patients after radiation therapy by comparing the incidence of unsatisfactory smear and the accuracy of detecting cervicovaginal lesions between the SurePath® and the conventional smear.

Patients and Methods: The investigators will invite all women who had received radiotherapy for cervical cancer in the investigators outpatient clinics. All enrolled cases will ask to receive randomly the SurePath® or the conventional smear.

Expected Results: The investigators will get the incidence of unsatisfactory smear and the accuracy of detecting cervicovaginal lesions between the SurePath® and the conventional smear in patients who underwent radiotherapy.

DETAILED DESCRIPTION:
Adequate specimen (specimen adequacy) is cervical or vaginal cytology single most important quality factors. 2001 Pap Bethesda System classification maintain its previous version, the Pap specimen is divided into satisfactory assessment and unsatisfactory evaluation two kinds; meet "satisfactory assessments "specimen standard, conventional Pap (conventional smear) requires at least 8,000-12,000-readable squamous cells, and liquid-based Pap (liquid-based smear) you need at least 5,000-readable squamous cell .

For squamous cell samples were determined to be adequate, yet to record their specimens have intrauterine neck or squamous transitional zone (transformation zone) border zone cells exist; quality indicators "Cell interpretation in part by inflammation or blood masking noise "of the specimen, if it can not be sentenced to 50-75% of epithelial cells can still be classified as read" satisfied "with the specimen, while more than 75% of the epithelial cells are obscured interference specimen is classified in the" unsatisfactory "specimen.

ELIGIBILITY:
Inclusion Criteria:

1. All women who had received radiotherapy for cervical cancer in our outpatient clinics.
2. Prior to joining test subjects for 90 days or more earlier had received a complete pelvic radiation therapy, including treatment of the cervix or vagina.
3. Subjects with radiation therapy (including combined chemical and radiation therapy or postoperative adjuvant [chemical] radiation therapy) for their first treatment.

Exclusion Criteria:

1. recurrence of cervical cancer
2. hormone treatment within 90 days
3. vaginal vault or cervix topical treatment within 90 days.
4. Subjects had or now have other malignancies

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With Cervical Cancer Receive Surepath for Screening | Women Receive Conventional Pap Smear for Screening
Started | 129 | 129
Completed | 129 | 129
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With Cervical Cancer Receive Surepath for Screening | Women Receive Conventional Pap Smear for Screening | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.44 (11.44) | 58.50 (8.13) | 57.97 (9.79)
Sex/Gender, Customized [Number; unit: participants] | 129 | 129 | 258

OUTCOME MEASURES:

1. Primary Outcome: the Percentage of Smears, That Were Difficulty in Making a Definite Diagnosis
Description: Comparing the percentage of smears, that were difficulty in making a definite diagnosis from smear owing to insufficient cells, between Surepath® and Conventional Smear in Women after Radiation Therapy for Cervical Cancer
Time Frame: 1 year
Population: Patients with cervical cancer who received radiation therapy
Measure: Number; unit: percentage of smears
Groups:
- Women Received Surepath for Screening: Women who received Surepath for screening the recurrence of cervical cancer.
- Women Received Conventional Pap Smear for Screening: Women who received conventional Pap smear for screening the recurrence of cervical cancer.
Arm/Group | Women Received Surepath for Screening | Women Received Conventional Pap Smear for Screening
Number analyzed (Participants) | 18 | 21
percentage of smears | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Women With Cervical Cancer Receive Surepath for Screening | Women Receive Conventional Pap Smear for Screening
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/129
Other Adverse Events (participants affected / at risk) | 0/129 | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes